CLINICAL TRIAL: NCT05145556
Title: Comparision of Direct Laryngoscopy and Video Laryngoscopy to Learn Successful Tracheal Intubation by Novices in Anaesthesiology
Brief Title: Teach Intubation by Novices in Anaesthesiology
Acronym: TeachIntub
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, PD Dr. med., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: JohannesGUIT
Record Dates: First submitted 2021-11-25; First posted 2021-12-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Learning Problem; Larynx
Keywords: Tracheal Intubation, Learning Technique, Laryngoscope
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Intervention Model Description: Starting with 100 tracheal intubations with conventional tracheal intubation and videolaryngoscopy and after 100 intubations change the device for the next 100 intubations
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscopy (McGrath Macintosh) (Experimental): First pass success rate using the videolaryngoscopy
  Interventions: Device: Videolarygoscopy
- conventional direct laryngoscopy (Experimental): First pass success rate using the conventional direct laryngoscopy
  Interventions: Device: conventional laryngoscopy

INTERVENTIONS:
Device: Videolarygoscopy — In a randomised order we evaluate the first pass success rate of the tracheal tube into the trachea.
  Arms: Videolaryngoscopy (McGrath Macintosh)
Device: conventional laryngoscopy — In a randomized order we evaluate the first pass success rate of the tracheal tube into the trachea.
  Arms: conventional direct laryngoscopy

SUMMARY:
Comparision of direct laryngoscopy and video laryngoscopy to learn successful tracheal intubation by novices in anaesthesiology

DETAILED DESCRIPTION:
Video laryngoscopy has been recommended as an alternative during difficult conventional direct laryngoscopy using the Macintosh blade. However, successful visualisation of the larynx and tracheal intubation using some of the indirect laryngoscopes or video laryngoscopy requires hand-eye coordination. To best of our knowledge in the current literature there are no data how is the best educative way to learn successful tracheal intubation by novices in anaesthesiology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* capacity to consent
* Present written informed consent of the research participant

Exclusion Criteria:

* Age <18 years
* Lack of consent
* inability to consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
First pass success rate | at intubation in 60 seconds
  successful tracheal intubation at the first attempt, compared to more than one attempt

SECONDARY OUTCOMES:
Time to ventilation | at intubation in 120 seconds
  From Insertion of the blase into the mouth until first ventilation
Cormack and Lehane Classification | at intubation in 120 seconds
  after insert the device the user describe the glottis visualisation
Overall success rate | at intubation in 120 seconds
  after two attempts using defined rescue techniques (e.g. rigid stylet, laryngeal mask)
Subjective Training Process | at one month
  after 25 intubation attempts

CONTACTS AND LOCATIONS:
Overall Officials: Marc MK Kriege, PD Dr, Principal Investigator — University JG, Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No